CLINICAL TRIAL: NCT07353359
Title: The Efficacy and Safety of Intranasal Negative Pressure Therapy (iNAP) in Patients With Mild Cognitive Impairment Complicated With Obstructive Sleep Apnea: A Randomized Controlled Trial
Brief Title: Effect of Intranasal Negative Pressure Therapy on Cognitive Function in Patients With Mild Cognitive Impairment and Obstructive Sleep Apnea
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025433; LinYanShen [2025] No.433-002 (Other: Xuanwu Hospital Capital Medical University)
Record Dates: First submitted 2026-01-09; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Mild Cognitive Impairment (MCI)
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iNAP group (Experimental): Participants use the iNAP device nightly for 24 weeks, combined with best support care.
  Interventions: Device: Intranasal Negative Pressure
- Control Group (No Intervention): Participants receive only sleep hygiene guidance without using the iNAP device.

INTERVENTIONS:
Device: Intranasal Negative Pressure — No interventions have been assigned to arm 'iNAP group' Intervention 'Intranasal Negative Pressure' has not been assigned to an arm/group.
  Arms: iNAP group

SUMMARY:
This study is a randomized controlled trial with two phases: pre-trial and formal trial. The pre-trial will include 5 participants to observe the 4-week adherence (≥4 hours/night) and safety (adverse event rate) of the iNAP device. For the formal trial, 60 patients with MCI and moderate-to-severe OSA will be stratified and block randomized (by baseline AHI levels: 15-30 events/h vs >30 events/h) into either the iNAP intervention group (using the device nightly for 24 weeks) or the control group (receiving only sleep hygiene guidance). The primary outcome is the change in MoCA scores from baseline at week 24. Secondary outcomes include AHI reduction rate, sleep efficiency, plasma Aβ42/Aβ40 ratio, cognitive assessments, and brain imaging indicators. Follow-up visits will occur at baseline, week 12, and week 24 to monitor cognitive function, sleep parameters, and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 50 and 75 years, regardless of gender.
2. Diagnosed with moderate-to-severe obstructive sleep apnea (OSA) via polysomnography (PSG), with an Apnea-Hypopnea Index (AHI) ≥ 15 events/hour.
3. Neuropsychological assessment consistent with mild cognitive impairment (MCI), defined as a Clinical Dementia Rating (CDR) of 0.5 and a Montreal Cognitive Assessment (MoCA) score between 20 and 26.
4. Successful completion of the iNAP device adaptation test (no significant oral discomfort, nausea, or other adverse reactions after 30 minutes of wear).
5. If using cognitive-enhancing medications (e.g., cholinesterase inhibitors, memantine), stable doses must be maintained for at least 12 weeks prior to baseline.
6. Voluntary signing of the informed consent form and willingness to comply with follow-up procedures.

Exclusion Criteria:

1. History of allergy to silicone components of the iNAP device. Severe nasal obstructive diseases (e.g., nasal polyps, moderate-to-severe chronic rhinitis) that impair nasal breathing function.
2. Acute cardio-cerebrovascular events (e.g., myocardial infarction, cerebral infarction) or acute exacerbation of moderate-to-severe lung diseases (e.g., COPD exacerbation) within the past 6 months.
3. Comorbidities with other sleep disorders (e.g., primary insomnia, narcolepsy, restless legs syndrome) that may interfere with OSA assessment.
4. Diagnosis of central nervous system diseases (e.g., epilepsy, sequelae of encephalitis) or severe mental illness (e.g., schizophrenia, major depression with SDS ≥ 63 points).
5. Severe aphasia or physical disability precluding completion of neuropsychological assessments.
6. Presence of consciousness disturbance from any cause.
7. Current diagnosis of depression or psychiatric disorders.
8. History of alcoholism, drug addiction, or neurological diseases known to cause cognitive impairment (e.g., traumatic brain injury, epilepsy, encephalitis, normal pressure hydrocephalus).
9. Concurrent participation in other clinical trials.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in MoCA Score from Baseline to Week 24 | Baseline (Day7～0 days) and Week 24 (Day 168±7 days)
  Montreal Cognitive Assessment (MoCA) scale ranges from 0 to 30, and higher value represents a better outcome. This study will use MoCA to assess changes in the global cognitive function after intervention.

SECONDARY OUTCOMES:
AHI Reduction Rate at Week 12 and Week 24 | Baseline, Week 12 (Day 84±7 days), and Week 24
  Percentage reduction in Apnea-Hypopnea Index (AHI) calculated as [(Baseline AHI - Follow-up AHI)/Baseline AHI] × 100%.
Change in Plasma Aβ42/Aβ40 Ratio | Baseline, Week 12, and Week 24
  Alteration in the ratio of plasma amyloid-beta 42 to 42/40
Change in Minimum Oxygen Saturation (LSaO₂) | Baseline, Week 12, and Week 24
  Increase in LSaO₂ from baseline, monitored via polysomnography (PSG)
Change in Sleep Efficiency | Baseline, Week 12, and Week 24
  Improvement in sleep efficiency [(Total Sleep Time/Time in Bed) × 100%] assessed by PSG.
Change in Auditory Verbal Learning Test Scores | Baseline, Week 12, and Week 24
  Auditory Verbal Learning Test (AVLT) scale ranges from 0 to 75 (sum of immediate recall and delayed recall), and higher value represents a better verbal memory. This study will use AVLT to assess changes in the episodic memory after intervention.
Changes in Plasma P-tau217 Concentrations | Baseline, Week 12, Week 24
  Reductions in plasma phosphorylated tau 217 (P-tau217) concentrations.
Changes in Structural MRI (sMRI) Metrics | Baseline, Week 12, Week 24
  Alterations in brain structure measured by T1-weighted sMRI.
Changes in Diffusion Tensor Imaging (DTI) Metrics | Baseline, Week 12, Week 24
  Improvements in white matter microstructural integrity and perivascular space (PVS) status.
Change in Resting-State fMRI (rs-fMRI) Brain Network Connectivity | Baseline, Week 12, Week 24
  Modifications in functional brain network connectivity compared to baseline.
Changes in EEG Metrics | Baseline, Week 12, Week 24
  Alterations in electroencephalogram (EEG) parameters (e.g., spectral power, coherence).
Changes in HAMA Score | Baseline, Week 12, Week 24
  Hamilton Anxiety Scale (HAMA) scale ranges from 0 to 56, and higher value represents more severe anxiety symptoms. This study will use HAMA to assess changes in the anxiety status after intervention.
Changes in HAMD Score | Baseline, Week 12, Week 24
  Hamilton Depression Scale (HAMD) scale ranges from 0 to 52, and higher value represents more severe depressive symptoms. This study will use HAMD to assess changes in the depressive status after intervention.
Incidence of Adverse Events (AEs) and Serious Adverse Events (SAEs) | Baseline, Week 12, Week 24
  Rate of treatment-related AEs (e.g., tongue soreness, increased salivation, dry mouth) and SAEs throughout the intervention period
change in Trail Making Test | Baseline, week 12, and week 24
  Trail Making Test (TMT) scale is quantified by completion time, and shorter time represents better executive function. This study will use TMT to assess changes in the cognitive flexibility and processing speed after intervention.
change in Stroop Color-Word Test | Baseline, week 12, and week 24
  Stroop Color-Word Test (SCWT) scale is quantified by interference score (reaction time of conflict trials minus reaction time of non-conflict trials), and smaller value represents better inhibitory control. This study will use SCWT to assess changes in the executive function after intervention.
Change in plasma Neurofilament Light Chain | baseline, week 12, and week 24
  alterations in plasma Neurofilament Light Chain concentrations
changes in plasma Glial Fibrillary Acidic Protein concentrations | baseline, week 12, and week 24
  changes in plasma Glial Fibrillary Acidic Protein concentrations

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No